CLINICAL TRIAL: NCT05746013
Title: Deciphering the Role of Dietary Fatty Acids on HDL Functionality
Brief Title: Lipoproteins and ImmunoMetabolism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Seville (Other)
Collaborators: Spanish National Research Council (Other Government)
Responsible Party: Principal Investigator, Sergio Montserrat de la Paz, Professor, University of Seville
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: US-1263458
Record Dates: First submitted 2022-11-17; First posted 2023-02-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2022-11

CONDITIONS: Obesity; Metabolic Syndrome; Metabolism Disorder; Inflammation; Immune System and Related Disorders
MeSH Terms: conditions — Obesity; Metabolic Syndrome; Metabolic Diseases; Inflammation | interventions — Fat Emulsions, Intravenous

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- No Fat meal (Placebo Comparator)
  Interventions: Dietary Supplement: Lipid Emulsion
- SFA meal (Experimental)
  Interventions: Dietary Supplement: Lipid Emulsion
- MUFA meal (Experimental)
  Interventions: Dietary Supplement: Lipid Emulsion
- PUFA meal (Experimental)
  Interventions: Dietary Supplement: Lipid Emulsion

INTERVENTIONS:
Dietary Supplement: Lipid Emulsion — The oral lipid emulsions will contain water, sucrose, emulsifier, flavouring, and the corresponding fat (50 g/m2 of body surface area): milk cream (SFA) or refined olive oil (MUFA) with or without a dose of omega-3 PUFA, which will consist of 920 mg of EPA and 760 mg of DHA.

SUMMARY:
Dietary interventions have been consistently proposed as a part of a comprehensive strategy to lower the incidence and severity of atherosclerosis and cardiovascular diseases (CVD). Excessive consumption of fats enriched in saturated fatty acids (SFA) is associated with an increased risk of atherosclerosis and other CVD. By contrast, replacement of SFA with monounsaturated fatty acids (MUFA) and omega-3 long-chain polyunsaturated fatty acids (ω-3 PUFA) has been reported to be inversely associated with risk of atherosclerosis. This is partly due to the ability of MUFA (and PUFA) in modulating low-density lipoprotein (LDL) and triglyceride-rich lipoprotein (TRL) lipid composition and oxidation status, and thereby the functionality of such lipoproteins. While most of the nutritional studies have focused on elucidating the mechanisms by which dietary fats affect LDL and TRL, little or nothing is known about the regulatory effect of MUFA and PUFA on structure and functional remodelling of high-density lipoproteins (HDL). There is clear evidence of an inverse association between plasma levels of HDL and the formation of atherosclerotic plaques. However, recent studies have suggested that HDL may not be as beneficial as thought at least in patients with established cardiometabolic disorders. In those patients, the HDL behaves as pro-inflammatory lipoproteins. Until now, few studies have addressed this "dark side" of HDL and has never been evaluated the role of dietary fatty acids on HDL plasticity (i.e. phenotype and functionality). A better understanding of this duality between anti-inflammatory and pro-inflammatory HDL would be relevant to prevent HDL-related atherogenic dyslipidemias and to provide personalized dietary advices for a successful management of atherogenic lipid profiles. This step of proof-of-principle will determine the instrumental role of major fatty acids present on a diet (SFA, MUFA and MUFA plus ω-3 PUFA) in promoting or reversing the phenotype of pro-inflammatory HDL. We expect to offer a novel insight on HDL and its relationship with dietary fatty acids through the following objectives: 1) To analyse acute changes in the lipidome, proteome and functional properties of HDL in humans (healthy volunteers and patients with metabolic syndrome) upon a challenge of a meal rich in SFA, MUFA or MUFA plus ω-3 PUFA; and 2) To analyse the influence of diets rich in SFA, MUFA and MUFA plus ω-3 PUFA on HDL plasticity in a preclinical animal model of diet-induced metabolic syndrome and that develops atherosclerosis.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of metabolic syndrome

Exclusion Criteria:

* Allergy to dairy products
* Allergy to fish oil
* Vegetarian
* Tobacco smoker
* Current or recent (<4 wk) use of fish oil supplements or more than four times fish/week
* Received innoculations within 2 mo of starting the study or planned to during the study
* Donated or intended to donate blood from 2 mo before the study till 2 mo after the study
* Unstable body weight (no weight gain/loss >3 kg)
* Medical condition that can interfere with the study outcome (i.e., biochemical evidence of active heart disease, renal impairment, hypothyroidism, liver dysfunction, etc.)
* Use of medications know to interfere with glucose homeostasis or lipid metabolism
* Use of anti-inflammatory medication, hormone or cytokine or growth factor therapies
* Abuse of drugs and/or alcohol
* Participation in another biomedical study within 1 mo before the first screening visit, or not wanting to be informed about chance-findings during screening.
* Severe diabetes, which requires application of insuin
* Diabetes-related complications.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Evolution of Glucose levels in postprandial state. | Up to 6 hours
  Blood glucose levels, measured by biochemical procedures (mg/dL).
Evolution of Insulin in postprandial state. | Up to 6 hours
  Blood Insulin levels, measured using ELISA procedures (pmol/L).
Evolution of C-peptide in postprandial state | Up to 6 hours
  C-peptide, using routine biochemical procedures (pmol/L).
Evolution of Trigliceride and NEFA parameters in postprandial state | Up to 6 hours
  Triglyceride and NEFA levels in plasma will be measured at several time-points postprandially using routine biochemical procedures (mg/dL)
Evolution of NAMPT in postprandial state | Up to 6 hours
  NAMP activity will be measured in plasma at several postprandial time-points using colorimetric techniques (UI/ml).
Evolution of cytokines in postprandial state | Up to 6 hours
  Pro-inflammatory and anti-inflammatory cytokines, including NFα, IL-1β, IL-6, IL-8, IL-10, ICAM-1, MCP-1, leptin, and adiponectin, in plasma will be measured using ELISA techniques (mg/dl).
Evolution of inflammatory markers in postprandial state. | Up to 6 hours
  The acute phase protein (hsCRP), PAI-1, fibrinogen, transferrin, albumin, and myeloperoxidase (MPO) will be measured using colorimetric techniques (mg/dl).
HDL lipoproteome | Up to 6 hours.
  HDL protein and lipid fractions HDL will be analysed by MALDI-TOF MS after employing an organic polymeric anion exchanger [Poly(GMA/EGDMA)] for lipoprotein enrichment from serum samples.
HDL antioxidant capacity | Up to 6 hours.
  HDL obtained from different postprandial points will be tested by their capacity to prevent LDL oxidation with an in vitro cell-free assay.
HDL cholesterol efflux capacity | Up to 6 hours.
  HDL cholesterol efflux capacity will be measured using fluorescent-labelled cholesterol. HDL extracted from serum at different postprandial points will be tested.
HDL LCAT activity | Up to 6 hours.
  Lecithin choltesteryl acyl transferase (LCAT) activity (UI/ml) of HDL obtained from different postprandial points will be measured using a fluorimetric cell-free assay.
HDL PON1 activity | Up to 6 hours
  Paraoxonse 1 (PON1) activity, of HDL obtained from serum at different postprandial tiems, will be measured using a colorimetric assay (pmol/mL).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Seville, Seville, Spain